CLINICAL TRIAL: NCT04590495
Title: The Effects of Cannabidiol on the Driving Ability of Healthy Adults: a Clinical Trial
Brief Title: The Effects of Cannabidiol on the Driving Ability of Healthy Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: West Virginia University (Other)
Responsible Party: Principal Investigator, Toni Marie Rudisill, Research Assistant Professor, West Virginia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2007073792
Record Dates: First submitted 2020-10-09; First posted 2020-10-19 (Actual); Results first posted 2022-09-15 (Actual); Last update posted 2022-09-15 (Actual); Status verified 2022-08

CONDITIONS: Driving Performance; Cognitive Impairment; Sedation Complication; Mood
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Cannabidiol; Oils

STUDY DESIGN:
Intervention Model Description: A randomized, parallel-group, double-blind, exploratory two-arm trial.
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- 300 mg Cannabidiol (CBD) oil (Active Comparator)
  Interventions: Drug: 300 mg Cannabidiol (CBD) oil
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: 300 mg Cannabidiol (CBD) oil — Participant will either be given a 300mg dosage of CBD oil. After consumption of the study drug, the participant will wait for 120 minutes to allow for digestion and for CBD to begin taking effect. Next, individuals will undergo a driving simulation and all participants will drive the same course. The simulator presents the individual with real life driving scenarios and is equipped with screens, a steering wheel, signals, and pedals. The participant will be instructed to drive the course for 25-35 minutes. They will be instructed to follow normal driving rules. The simulation will include highway, suburban, rural, and urban driving scenarios which will incorporate turns, changes in speed, and avoidance of cars/pedestrians.
  Arms: 300 mg Cannabidiol (CBD) oil
Drug: Placebo — Participant will either be given a placebo . After consumption of the study drug, the participant will wait for 120 minutes to allow for digestion and for CBD to begin taking effect. Next, individuals will undergo a driving simulation and all participants will drive the same course. The simulator presents the individual with real life driving scenarios and is equipped with screens, a steering wheel, signals, and pedals. The participant will be instructed to drive the course for 25-35 minutes. They will be instructed to follow normal driving rules. The simulation will include highway, suburban, rural, and urban driving scenarios which will incorporate turns, changes in speed, and avoidance of cars/pedestrians.
  Arms: Placebo

SUMMARY:
A randomized, parallel-group, double-blind, exploratory two-arm trial to assess the effects of CBD on driving ability along with changes in psychological status (i.e. mood, drowsiness, sedation) and cognitive function. Forty healthy West Virginia University (WVU) students will be allocated and randomized to receive: (1) 300 mg of pure CBD oil or (N=20) (2) placebo matched in appearance and taste (N=20). After consuming the study drug, each individual will participate in a 25-35-minute driving simulation and their driving performance measured. To assess changes in psychological status (i.e. mood, drowsiness, sedation) and drug impairment-related cognitive function, the Visual Analog Mood Scale, Stanford Sleepiness Scale , Digital Symbol Substitution Test, Trail Making Test Part A and B, Psychomotor Vigilance Test, and Simple Reaction Time test will also be administered to participants at baseline (prior to study drug consumption) and following completion of the driving simulation test. The entire protocol will be completed in one day and should take 4-4.5 hours to complete for each participant.

ELIGIBILITY:
Inclusion Criteria:

1) the participant must be currently enrolled as a WVU student, 2) be 18-30 years of age at time of study, 3) have a current drivers' license issued from any state in the United States, 4) has driven at least once in the past 30 days 5) is able to speak and read English, 6) is willing to be randomized and comply with study requirements including a urine drug test on the day they consent to participate in the experiment and complete a test drive to ensure the absence of simulation sickness, 7) not currently taking any daily prescription medications other than birth control, 8) have not been diagnosed with any serious chronic disease by a licensed healthcare provider (including but not limited to Alzheimer's and related dementias, Parkinson's disease or other neurodegenerative disorder, major depressive or anxiety disorder, schizophrenia or other serious mental illness, arrhythmias, cataracts, glaucoma, chronic obstructive pulmonary disease, diabetes, epilepsy, sleep apnea, and fibromyalgia), and 9) has an individual able to drive them home after testing or is willing to be driven home by study staff after testing completion.

Exclusion Criteria:

Participants will be excluded if they 1) currently smoke or use tobacco products, 2) have used illegal drugs (including cocaine/crack, heroin, methamphetamine, 3,4-methylenedioxy-methamphetamine, inhalants, phencyclidine, lysergic acid, mushrooms, or marijuana) in the past 30 days, 3) has consumed CBD in the past 7 days, or 4) is currently pregnant or lactating

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2021-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Toni Marie Rudisill, MS, PhD, Principal Investigator — West Virginia University
Locations (1):
- West Virginia University, Morgantown, West Virginia, United States

IPD SHARING:
Plan to Share IPD: No
We do not plan to share these data.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study took place at West Virginia University in Morgantown, West Virginia. Participants were recruited from April 1, 2021 until Dec 1, 2021 when the target enrollment was met.
Period: Overall Study
Arm/Group | 300 mg Cannabidiol (CBD) Oil | Placebo
Started | 21 | 19
Completed | 21 | 19
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 300 mg Cannabidiol (CBD) Oil | Placebo | Total
Number analyzed (Participants) | 21 | 19 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 21.4 (2.8) | 21.0 (2.7) | 21.2 (2.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 10 | 21
  Male | 10 | 9 | 19
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 18 | 16 | 34
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 3 | 6
Body mass index [Mean (Standard Deviation); unit: Kilogram/meters squared] | 26.3 (6.3) | 25.6 (3.6) | 26.0 (5.2)
West Virginia Residency [Count of Participants; unit: Participants]
  West Virginia Resident | 12 | 13 | 25
  Non West Virginia Resident | 9 | 6 | 15
Undergraduate student status [Count of Participants; unit: Participants]
  Undergraduate Student | 13 | 15 | 28
  Graduate Student | 8 | 4 | 12
Employment status [Count of Participants; unit: Participants]
  Employed | 11 | 10 | 21
  Not employed | 10 | 9 | 19
Number of hours spent playing video games [Mean (Standard Deviation); unit: Hours] | 5.6 (5.1) | 8.6 (13.8) | 7.1 (10.2)
Miles driven per week [Mean (Standard Deviation); unit: miles/week] | 49.9 (60.5) | 48.9 (43.7) | 49.5 (52.7)
Hours of sleep previous night [Mean (Standard Deviation); unit: Hours] | 7.3 (1.0) | 7.1 (1.2) | 7.2 (1.1)
Average daily caffeine consumption [Mean (Standard Deviation); unit: ounces] | 12.9 (13.1) | 10.1 (9.8) | 11.5 (11.5)
Ever used cannabidiol previously [Count of Participants; unit: Participants]
  Used Cannabidiol previously | 4 | 5 | 9
  Did not use Cannabidiol previously | 17 | 14 | 31

OUTCOME MEASURES:

1. Primary Outcome: Driving Performance - Percent of Time Spent Out of Lane
Description: From driving simulation. A greater percentage of time spent driving out of lane indicates worse performance. Min=0 max=100%
Time Frame: 1.5 hour post intervention
Measure: Mean (Standard Deviation); unit: Percent time spent driving out of lane
Arm/Group | 300 mg Cannabidiol (CBD) Oil | Placebo
Number analyzed (Participants) | 21 | 19
Percent time spent driving out of lane | 4.41 (2.44) | 4.34 (2.09)
Statistical Analysis 1: Comparison: Placebo; Test type: Superiority; p = 0.9460, Mann Whitney U Test

2. Primary Outcome: Driving Performance - Number of Collisions.
Description: From driving simulation. A greater number of collisions indicate worse performance. Min=0 max=infinity
Time Frame: 1.5 hour post intervention
Measure: Mean (Standard Deviation); unit: Number of collisions
Arm/Group | 300 mg Cannabidiol (CBD) Oil | Placebo
Number analyzed (Participants) | 21 | 19
Number of collisions | 0.90 (1.09) | 0.68 (0.95)
Statistical Analysis 1: Comparison: Placebo; Test type: Superiority; p = 0.5699, Mann Whitney U Test

3. Primary Outcome: Driving Performance - Brake Reaction Time
Description: Mean reaction time to stimuli from driving simulation. Longer reaction times indicate worst performance. Min=0 max=infinity
Time Frame: 1.5 hour post intervention
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | 300 mg Cannabidiol (CBD) Oil | Placebo
Number analyzed (Participants) | 21 | 19
Seconds | 0.60 (0.11) | 0.58 (0.12)
Statistical Analysis 1: Comparison: Placebo; Test type: Superiority; p = 0.6068, t-test, 2 sided

4. Primary Outcome: Driving Performance - Lateral Position in Lane
Description: Mean standard deviation of lateral position in lane under consistent speed from driving simulation. Larger standard deviations in lane position indicate worse performance. Min=0 max=infinity
Time Frame: 1.5 hour post intervention
Measure: Mean (Standard Deviation); unit: Feet
Arm/Group | 300 mg Cannabidiol (CBD) Oil | Placebo
Number analyzed (Participants) | 21 | 19
Feet | 4.37 (2.22) | 3.88 (2.49)
Statistical Analysis 1: Comparison: Placebo; Test type: Superiority; p = 0.9030, Mann Whitney U Test

5. Primary Outcome: Driving Performance-percent of Time Spent Driving Above Speed Limit
Description: From driving simulation. This is the percent of drive time that the driver spent driving above the speed limit. Greater percentage indicates worse performance.
Time Frame: 1.5 hour post intervention
Measure: Mean (Standard Deviation); unit: Percent time driving over speed limit
Arm/Group | 300 mg Cannabidiol (CBD) Oil | Placebo
Number analyzed (Participants) | 21 | 19
Percent time driving over speed limit | 5.83 (6.02) | 8.27 (9.58)
Statistical Analysis 1: Comparison: Placebo; Test type: Superiority; p = 0.2668, t-test, 2 sided

6. Secondary Outcome: Change in Baseline VAMS for Mental Sedation
Description: Visual Analog Mood Scale (VAMS). Mental sedation: sum of scores from questions 1, 4, 11, 13 on VAMS - higher scores indicate more mental sedation. Total min=0 Total max=400
Time Frame: 4 hours after baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 300 mg Cannabidiol (CBD) Oil | Placebo
Number analyzed (Participants) | 21 | 19
score on a scale | 148.7 (80.1) | 161.3 (78.3)
Statistical Analysis 1: Comparison: Placebo; Test type: Superiority; p = 0.8749, paired t test — adjusted for baseline VAMS score

7. Secondary Outcome: Change in Baseline VAMS--Physical Sedation
Description: Visual Analog Mood Scale (VAMS). Physical sedation: sum of scores from questions 3, 5, 6, 16 on VAMS - higher scores indicate more physical sedation. Total min=0 Total max=400
Time Frame: 4 hours after baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 300 mg Cannabidiol (CBD) Oil | Placebo
Number analyzed (Participants) | 21 | 19
score on a scale | 135.6 (65.3) | 152.7 (71.0)
Statistical Analysis 1: Comparison: Placebo; Test type: Superiority; p = 0.7922, paired t test — adjusted for baseline VAMS score for physical sedation

8. Secondary Outcome: Change in Baseline SSS
Description: Stanford Sleepiness Scale (SSS). Self-reported sleepiness, The SSS is a Likert-type scale which assess mental and physical sedation and sleepiness, respectively, at that moment and time. SSS only consists of 1 question that is scaled from 1 to 7, with 7 being a higher or worse score (i.e. more sleepy and sedated)
Time Frame: 4 hours after baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 300 mg Cannabidiol (CBD) Oil | Placebo
Number analyzed (Participants) | 21 | 19
units on a scale | 2.67 (1.32) | 2.63 (1.42)
Statistical Analysis 1: Comparison: Placebo; Test type: Superiority; p = 0.9925, paired t test — adjusted for baseline SSS score

9. Secondary Outcome: Change in Baseline TMT Part A
Description: Trail Making Test (TMT). Time to accurately complete Part A . The TMT measures executive function and consists of two parts; the first part requires participants to connect numbers in ascending order, while the second part requires individuals to connect numbers and letters in sequence. The test is scored by the time it takes to accurately complete each test. Increases in time correlate with greater impairment.
Time Frame: 4 hours after baseline
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | 300 mg Cannabidiol (CBD) Oil | Placebo
Number analyzed (Participants) | 21 | 19
Seconds | 14.2 (4.1) | 15.6 (5.2)
Statistical Analysis 1: Comparison: Placebo; Test type: Superiority; p = 0.2628, paired t test — adjusted for baseline score

10. Secondary Outcome: Change in Baseline TMT Part B
Description: Trail Making Test (TMT). Time to accurately complete Part B. The TMT measures executive function and consists of two parts; the first part requires participants to connect numbers in ascending order, while the second part requires individuals to connect numbers and letters in sequence. The test is scored by the time it takes to accurately complete each test. Increases in time correlate with greater impairment.
Time Frame: 4 hours after baseline
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | 300 mg Cannabidiol (CBD) Oil | Placebo
Number analyzed (Participants) | 21 | 19
Seconds | 29.7 (8.9) | 37.1 (15.9)
Statistical Analysis 1: Comparison: Placebo; Test type: Superiority; p = 0.0347, paired t test — adjusted for baseline scores

11. Secondary Outcome: Change in Baseline DSST
Description: Digital Symbol Substitution Test (DSST). Number of correct symbols completed within 60 seconds. The test is scored by the degree of completion and accuracy over a timed 60 second period. More accurate completion (i.e. higher the score) indicates better cognitive functioning. Min=0 Max=90
Time Frame: 4 hours after baseline
Measure: Mean (Standard Deviation); unit: Number of correct symbols
Arm/Group | 300 mg Cannabidiol (CBD) Oil | Placebo
Number analyzed (Participants) | 21 | 19
Number of correct symbols | 74.5 (8.1) | 71.8 (12.1)
Statistical Analysis 1: Comparison: Placebo; Test type: Superiority; p = 0.6331, paired t test — adjusted for baseline score

12. Secondary Outcome: Change in Baseline PVT
Description: Psychomotor Vigilance Test (PVT). Mean reaction time (in milliseconds) when responding to a stimuli that appears on a computer screen. Longer reaction time means worse vigilance. Min=0 max=infinity
Time Frame: 4 hours after baseline
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | 300 mg Cannabidiol (CBD) Oil | Placebo
Number analyzed (Participants) | 21 | 19
milliseconds | 331.7 (37.7) | 330.0 (32.7)
Statistical Analysis 1: Comparison: Placebo; Test type: Superiority; p = 0.4720, paired t test — adjusted for baseline score

13. Secondary Outcome: Change in Baseline SRT for Sound #1
Description: Simple Reaction Time test (SRT). Mean reaction time to stimuli that appears on a computer screen. Longer reaction times mean a decrease in reaction time. Min=0 max=infinity. Two separate sounds were emitted. Data were obtained for participants reaction to each separate sound
Time Frame: 4 hours after baseline
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | 300 mg Cannabidiol (CBD) Oil | Placebo
Number analyzed (Participants) | 21 | 19
milliseconds | 241.4 (22.1) | 244.6 (30.2)
Statistical Analysis 1: Comparison: Placebo; Test type: Superiority; p = 0.0200, paired t test — adjusted for baseline reaction time

14. Secondary Outcome: Change in Baseline SRT--sound #2
Description: as for outcome 13
Time Frame: 4 hours after baseline
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | 300 mg Cannabidiol (CBD) Oil | Placebo
Number analyzed (Participants) | 21 | 19
milliseconds | 239.6 (20.8) | 240.4 (48.0)
Statistical Analysis 1: Comparison: Placebo; Test type: Superiority; p = 0.0620, paired t test — adjusted for baseline reaction time

ADVERSE EVENTS:
Time Frame: As the half life of cannabidiol is ~17 hours, all participants were contacted via cellphone 8-12 hours and ~24 hours post-testing to inquire about adverse events. These conversations and potential adverse events were logged by study staff in an electronic survey.
Arm/Group | 300 mg Cannabidiol (CBD) Oil | Placebo
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/19
Other Adverse Events (participants affected / at risk) | 0/21 | 0/19

LIMITATIONS AND CAVEATS:
Only one dosage of CBD was utilized, and this dose may not reflect "normal" use of CBD. Participants were recruited from a university so results may not be generalizable to the general population. Previous studies have shown that CBD's max absorption occurs 2-5 hours post-consumption. To balance participant burden, a two-hour waiting period between dosing and simulation was chosen. It is possible that max absorption and full effect of the drug was not reached amongst some participants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2021-09-27): https://cdn.clinicaltrials.gov/large-docs/95/NCT04590495/Prot_SAP_ICF_000.pdf